CLINICAL TRIAL: NCT00169260
Title: Proactive Cessation Intervention With Biomarker Feedback
Brief Title: Proactive Health Intervention for Tobacco Users (Get PHIT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CA100341-02 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Smoking
Keywords: smoking; tobacco; behavior therapy
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention
  Interventions: Behavioral: motivational counseling
- 2 (Placebo Comparator): Control
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: motivational counseling — behavioral motivational counselling
  Arms: 1
Behavioral: placebo
  Arms: 2

SUMMARY:
The goal of this study is to understand how information about smokers' health risks affects their attitudes, mood, and behavior.

DETAILED DESCRIPTION:
The current study will test a community-based, tobacco intervention. The project will compare the effects of a proactive, personally-tailored, biologically-based motivational intervention to those of a proactive, generic motivational intervention for smoking cessation. The biologically-based motivational treatment will include feedback on participants' carbon monoxide (CO) exposure (expired CO and estimated carboxyhemoglobin levels), pulmonary functioning assessed via spirometry, and self-reported smoking-related symptoms. All participants will be given equal access to action-oriented treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old,
* smoke greater than or equal to 15 cigarettes a day,
* have an expired CO level greater than or equal to 10 ppm,
* are not currently being treated for smoking cessation,
* can read and write in English,
* provide contact information,
* agree to the study requirements,
* have no medical contraindications for spirometry assessment,
* and no an obvious cognitive or physical impairment that would preclude their ability to comprehend or fully participate in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2005-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Motivation to quit smoking, utilization of available resources, smoking cessation rate | 1 year

SECONDARY OUTCOMES:
Measurement of emotional distress, and mediators/moderators of primary outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B McClure, Ph.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] McClure JB, Ludman EJ, Grothaus L, Pabiniak C, Richards J. Impact of spirometry feedback and brief motivational counseling on long-term smoking outcomes: a comparison of smokers with and without lung impairment. Patient Educ Couns. 2010 Aug;80(2):280-3. doi: 10.1016/j.pec.2009.11.002. PMID 20434863
- [Derived] McClure JB, Ludman EJ, Grothaus L, Pabiniak C, Richards J. Impact of a brief motivational smoking cessation intervention the Get PHIT randomized controlled trial. Am J Prev Med. 2009 Aug;37(2):116-23. doi: 10.1016/j.amepre.2009.03.018. Epub 2009 Jun 12. PMID 19524389